CLINICAL TRIAL: NCT00679705
Title: Pilot Study: A Dose-Response Finding Study of Ritodrine (Pre-Par®) to Find the Highest Well Tolerated Dose in Young, Healthy, Female Volunteers. To Find the Size-Order of the Hemodynamical Effects of Ritodrine (PrePar®) and Atosiban (Tractocile®) to Determine the Relevance of a PK/PD-Modelling in the Final Study. Final Study: Investigating the Influence of Tocolytical Medications: Ritodrine (PrePar®) and Atosiban (Tractocile®) at the Clinical Dose on the Hemodynamics and Arterial Function in Healthy Female Volunteers, Compared to Placebo During Continuous Intravenous Infusion.
Brief Title: Influence of Tocolytical Medications on Hemodynamics (Central and Peripheral) and Vascular Function in a Pilot Study to Determine the Design of the Final Study and the Final Study Itself
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Luc Van Bortel, MD, PhD, University Hospital Ghent
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/110
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Hemodynamics and arterial function of healthy females
MeSH Terms: interventions — Ritodrine; atosiban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Ritodrine (Pre-Par)
  Interventions: Drug: Ritodrine
- 2 (Experimental): Atosiban (Tractocile)
  Interventions: Drug: Atosiban
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritodrine — Ritodrine (Pre-Par), maximum 400 µg/minute, IV
  Arms: 1
Drug: Atosiban — Atosiban (Tractocile), maximum 300 µg/minute, IV
  Arms: 2
Drug: Placebo — Glucose 5%, IV
  Arms: 3

SUMMARY:
This trial will consist of two parts:

A pilot study in a three-way cross over trial to determine the highest well tolerated dose of Ritodrine (Pre-Par®), the impact of Atosiban (Tractocile®) on the hemodynamics and hence the design of the final study.

The final study is planned as a three-way crossover trial to investigate and compare the cardiovascular effects of Ritodrine, Atosiban and placebo to relate those effects to the pharmacokinetics of Ritodrine and Atosiban (PK/PD modelling).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40 years old;
* In good health, especially no cardiovascular diseases, obstructive lung diseases, chronic kidney diseases or diabetes mellitus.
* Using a proper anticonception method (orally, subcutaneously);
* A negative pregnancy test.

Exclusion Criteria:

* Intolerance of Ritodrine;
* On chronic medication, except oral and subcutaneous contraception
* History or present presentation of cardiac arrythmias;
* Risk of being pregnant or less than 6 months postpartum;
* Giving breastfeeding;
* Previous uteral surgery;
* Using an intra-uteral device (IUD);
* A severe addiction: nicotine (> 10 cigarettes/day), alcohol (> 3 units/day), caffeine (> 5 units/day) or any extralegally drugs.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Hemodynamical effects of Ritodrine and Atosiban in comparison of those of placebo. | 240 minutes

SECONDARY OUTCOMES:
Effect of the specific dosing levels of the medications on the level of arterial stiffness | 240 minutes
Effect of the specific dosing levels of the medications on the effects of the peripheral pulse wave reflections on the central, systolic blood pressure | 240 minutes
Effect of the specific dosing levels of the medications on the distensibility of the blood vessel wall | 240 minutes
Effect of the specific dosing levels of the medications on the cardiac output and total peripheral resistance | 240 minutes
Effect of the specific dosing levels of the medications on peripheral brachial, systolic and diastolic blood pressure | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Bortel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be